CLINICAL TRIAL: NCT03584360
Title: Study Role of the Local Treatments on the Microbiome Modulation in the Psoriatic Skin. Study Monocentric, Interventional, Randomized and Single-blind
Brief Title: Role of Topical Treatments in the Modulation of Skin Microbiome in Psoriatic Skin
Acronym: Microbiome&Pso
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-PP-03
Record Dates: First submitted 2018-06-18; First posted 2018-07-12 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Intervention Model Description: patients apply different treatment to two areas with psoriasis
Who Masked: Investigator
Masking Description: The patient will not say the treatment he puts on each treatment area
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- betamethasone-calcipotriol versus placebo (Experimental): In this arm we will compared the application association of betamethasone-calcipotriol foam in an area versus a placebo foam in an other area during 4 weeks.
  Interventions: Drug: Betamethasone-Calcipotriene Topical
- betamethasone-calcipotriol versus betamethasone (Experimental): In this arm we will compared the application association of betamethasone-calcipotriol foam in an area versus a betamethasone pomade in an other area during 4 weeks.
  Interventions: Drug: Betamethasone-Calcipotriene Topical
- betamethasone-calcipotriol versus propionate of clobetasol (Experimental): In this arm we will compared the application association of betamethasone-calcipotriol foam in an area versus a propionate of clobetasol pomade in an other area during 4 weeks.
  Interventions: Drug: Betamethasone-Calcipotriene Topical

INTERVENTIONS:
Drug: Betamethasone-Calcipotriene Topical — Comparison between betamethasone-calcipotriol and placebo
  Arms: betamethasone-calcipotriol versus placebo
Drug: Betamethasone-Calcipotriene Topical — Comparison between betamethasone-calcipotriol and betamethasone
  Arms: betamethasone-calcipotriol versus betamethasone
Drug: Betamethasone-Calcipotriene Topical — Comparison between betamethasone-calcipotriol and propionate de clobetasol
  Arms: betamethasone-calcipotriol versus propionate of clobetasol

SUMMARY:
Changes in microbiome have been reported recently in psoriasis lesions compared to healthy surround skin. Preliminary data showed that systemic treatments of psoriasis induce modification of the skin microbiome that becomes similar to healthy individuals after successful treatment. The causative role of microbiome in psoriasis remains in debate. The modification of skin microbiome is suspected to be able to activate the innate immune response, namely natural killers (NKs) and immune lymphoid cells (ILCs). Three types of ILCs have been reported. ILC1 (immune lymphoid cells1) that trigger a Th1 response, ILC2 (immune lymphoid cells 2) that stimulate Th2 response and ILC3 (immune lymphoid cells 3) that induce Th17 response. Interestingly, ILC2 have been reported to be increased in atopic dermatitis while ILC3 are increased in psoriasis.

DETAILED DESCRIPTION:
To date, there is no data on the impact of topical treatments in skin microbiome and in innate cells in psoriasis lesions. However, topical treatments remain in most cases the first and the more widely used option for mild psoriasis which represent the more prevalent form of psoriasis. Thus, it appears of great interest to assess the effect of topical psoriasis treatments on skin microbiome. To this respect, topical steroids by their action both on the inflammation but also potentially on bacteria are suspected to induce potent changes in the microbiome in treated psoriasis lesions. calcipotriol has been demonstrated to have a beneficial effect on psoriasis thanks to its action on keratinocyte differentiation and its combination with topical steroids has been shown to be superior in treating psoriasis as compared to topical steroids alone. It could be hypothesized that calcipotriol could also modify the skin microbiome.

The main objective of this study intra individual prospective study is to compare the respective effect of betamethasone associated with calcipotriol foam and placebo foam in one hand and betamethasone with calcipotriol foam to betamethasone ointment on the other hand, on skin microbiome after 4 weeks of treatments on knee or elbow lesions.

Secondary objectives are to study the impact of the treatments on ILCs (numbers and relative proportion in the 3 types) and NK in the lesions and their potential correlation with the modification of the microbiome (of note ILC can be detected and characterized in situ in skin.) To compare the relative effectiveness of the two products on targets psoriasis lesions. Tolerance and potential side effects will be also studied.

Main endpoint: quantitative and qualitative assessment of microbes on psoriasis lesions before and after the treatments compared to surrounding healthy skin control.

Secondary endpoints: Presence and types of ILCs and NK in the lesional psoriatic skin before and after treatment compared with control healthy skin assessed using immunohistofluorescence. Targeted PASI or PGA (physician Global Assessment) for the efficacy. Potential side effects.

Patients: 30 with mild psoriasis (PASI <10) affecting elbows and knees in a symmetrical manner aged of at least 18.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age who have signed and dated an informed information and consent form,
* Subject presenting psoriasis vulgaris with lesions symmetrical in size and severity, localized on the elbows and the knees and having a severity score (PASI) <=10. The lesions must have an area of at least 4 cm²,

Exclusion Criteria:

* Psoriasis in gout, erythrodermic, exfoliative or pustular
* Subject who has received systemic treatment and has a potential action on psoriasis vulgaris
* Subject who received topical treatments or neutral emollients within 4 weeks
* Subject who received antibiotic treatment in the three months preceding the randomization visit
* Subject with known or suspected hypersensitivity to any of the constituents of the products in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Quantitative evaluation of bacterial microbiota on psoriasis lesions and surrounding healthy skin by 16S rRNA (ribosomal ribonucleic acid 16S) amplification coupled with high throughput sequencing | after 4 weeks of treatment
Qualitative evaluation of bacterial microbiota on psoriasis lesions and surrounding healthy skin by 16S rRNA (ribosomal ribonucleic acid 16S) amplification coupled with high throughput sequencing | after 4 weeks of treatment

SECONDARY OUTCOMES:
Targetted Psoriasis Area and Severity Index for the effectiveness of the products tested. | after 4 weeks of treatment
  Evaluated by PASI score (PASI= Psoriasis Area Severity Index) minimum = 0 = Absence of psoriasis maximum = 4 = very severe psoriasis
Number of ILCs and NKs on skin biopsies using immunohistochemistry | after 4 weeks of treatment
Types of ILCs and NKs on skin biopsies using immunohistochemistry | after 4 weeks of treatment
Score of overall evaluation of the investigator's treatment | after 4 weeks of treatment
  Evaluated by physician global assessment (PGA) score PGA = physician global assessment minimum = 0 = healing maximum = 5 = very severe psoriasis
Evaluation of tolerance | after 4 weeks of treatment
  evaluated numbers of serious adverse events
Occurrence of possible adverse effects | after 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PASSERON, MD, PhD, Principal Investigator — university hospital center of nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Javitz HS, Ward MM, Farber E, Nail L, Vallow SG. The direct cost of care for psoriasis and psoriatic arthritis in the United States. J Am Acad Dermatol. 2002 Jun;46(6):850-60. doi: 10.1067/mjd.2002.119669. PMID 12063481
- [Background] Schmitt JM, Ford DE. Work limitations and productivity loss are associated with health-related quality of life but not with clinical severity in patients with psoriasis. Dermatology. 2006;213(2):102-10. doi: 10.1159/000093848. PMID 16902286
- [Background] Wong VW, Martindale RG, Longaker MT, Gurtner GC. From germ theory to germ therapy: skin microbiota, chronic wounds, and probiotics. Plast Reconstr Surg. 2013 Nov;132(5):854e-861e. doi: 10.1097/PRS.0b013e3182a3c11e. PMID 24165637
- [Background] Mathieu A, Vogel TM, Simonet P. The future of skin metagenomics. Res Microbiol. 2014 Feb-Mar;165(2):69-76. doi: 10.1016/j.resmic.2013.12.002. Epub 2013 Dec 20. PMID 24361423
- [Background] Kong HH, Andersson B, Clavel T, Common JE, Jackson SA, Olson ND, Segre JA, Traidl-Hoffmann C. Performing Skin Microbiome Research: A Method to the Madness. J Invest Dermatol. 2017 Mar;137(3):561-568. doi: 10.1016/j.jid.2016.10.033. Epub 2017 Jan 4. PMID 28063650
- [Background] Kong HH, Segre JA. The Molecular Revolution in Cutaneous Biology: Investigating the Skin Microbiome. J Invest Dermatol. 2017 May;137(5):e119-e122. doi: 10.1016/j.jid.2016.07.045. PMID 28411842
- [Result] Naldi L, Svensson A, Diepgen T, Elsner P, Grob JJ, Coenraads PJ, Bavinck JN, Williams H; European Dermato-Epidemiology Network. Randomized clinical trials for psoriasis 1977-2000: the EDEN survey. J Invest Dermatol. 2003 May;120(5):738-41. doi: 10.1046/j.1523-1747.2003.12145.x. PMID 12713574